CLINICAL TRIAL: NCT03116607
Title: Impact of a Pharmaceutical Intervention Program at Readmission and User Satisfaction in a Emergency Department, Randomized Clinical Study
Brief Title: Pharmaceutical Intervention Program at Readmission and User Satisfaction in a Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Matías Fernando Martínez Olguín, Pharmacist, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCh2015
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Personal Satisfaction
Keywords: User satisfaction; Readmission; Emergency department; Pharmaceutical intervention
MeSH Terms: conditions — Personal Satisfaction; Emergencies | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: parallels groups: control arm will recieve normal healthcare, intervention arm will recieve a pharmaceutilcal intervention program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive the usual hospital care. In addition, an interview that allows the characterization of the sample and the measurement of variables such as adherence, problems related to medication and user satisfaction.
- Intervened (Experimental): The intervention group will receive a Pharmaceutical Intervention Program during their stay in the Service and discharge.
  In addition, an interview that allows the characterization of the sample and the measurement of variables such as adherence, problems related to medication and user satisfaction.
  patient education/ recommendations to the health team
  Interventions: Other: patient education/ recommendations to the health team

INTERVENTIONS:
Other: patient education/ recommendations to the health team — The intervention group will receive a Pharmaceutical Intervention Program during their stay in the Service and discharge that includes an analysis of the therapy indicated by the physician, evaluating the safer alternatives for the type of patient and the special conditions of their pathology, with emphasis on Assessments of effectiveness, safety and tolerability of medication, drug interactions, possible adverse events, dose adjustments as necessary according to patient conditions; Verification that the administration is optimal, including the choice of the best route for this and the time in which the drugs are infused to the patient.
  Arms: Intervened

SUMMARY:
A randomized clinical trial with two parallel groups (control and intervened) in the Emergency Department (ED) at the Clinical Hospital of the University of Chile will take place. The sample will be of 996 patients (498 per group).

The control group will receive hospital care and discharge plan usual, while the intervention group also receive a Program of Pharmaceutical Interventions while in the service and at discharge, which includes an analysis of the therapy recommended by the physician, assessing the safer alternatives for the patient population and the special conditions of their pathology, emphasizing evaluations of effectiveness, safety and tolerability of medication, drug interactions, potential adverse events, dose adjustments as needed according to the patient's condition ; verification that the administration is optimal, including choosing the best route to this and the time when the drugs are infused into the patient.Interventions aimed at patient occur during the stay and at discharge, focusing on clarifying administration regimens, reasons for using drugs, prevent drug-related problems, clarify doubts and educate about pharmacotherapy and make a reinforcement of adherence.

The selection and patient recruitment will take place during the first hour of admission to care box, where they were invited to participate and signed informed consent.

In both groups, a doctor and a pharmacist, blind to treatment assignment, will gather information during the stay, discharge and post-discharge, the latter by telephone 30 days after discharge from the ED, in this second interview also verify the existence of a readmission and / or unscheduled medical consultation. In addition, discharge of each patient satisfaction was measured with respect to the service received by a user satisfaction survey applied by external and impartial staff. In addition, two independent trained evaluators (Emergency Medical and Pharmaceutical Chemistry), blinded to treatment assignment, evaluate the background of each case and by consensus allocated the presence of problems related to drugs, and classified as preventable or not preventable, according severity.

X2 test or Fisher exact test was used to test the hypothesis that the Programme of Pharmaceutical Interventions decreases at least 30% the user dissatisfaction compared with usual care in the ED.

DETAILED DESCRIPTION:
Process:

For the selection of patients, a research team consisting of a Physician and a Pharmaceutical Chemist review the inclusion and exclusion criteria within the first hour after the patient enters the care box. Patients who meet the selection criteria are invited to participate in the study and sign the informed consent form. To standardize the sampling and avoid differences by daily or seasonal variation are included in the study of 6 patients per day.

For each of the included patients, information will be collected that allows the characterization: sociodemographic, which includes: sex, age, foresight, schooling, marital status; Morbid antecedents before, during the care and after the high diagnostic illness, reason of admission and previous hospitalizations; Pharmacotherapeutic which includes medicines used, dosage, self-medication, adherence (Morisky & Green Scale), performed before, during the stay in the emergency department and high and post discharge. In addition, the Triage category and the duration of the stay are recorded.

In both groups, a physician and a pharmacist, blind to the allocation of treatment, collect the demographic, morbid and pharmacotherapeutic antecedents, by means of a file specially designed for the study. The post-discharge evaluation is done through the telephone interview 30 days after the discharge from the US.

All information collected on the follow-up sheets of each study patient will be added to an Excel® database. A project investigator will be responsible for ensuring the monitoring of the study, ensuring that Good Clinical Practices are complied with, as well as the quality and reliability of the information recorded on both the records and the database. Both the database and each of the study collection records will include only a patient identification code, in order to maintain their confidentiality. The list that relates the code to the patient's name will be kept protected with access only to the principal investigator.

In the case of the patients who are part of the intervention group, in addition to the care received by the control group, I received a pharmaceutical care program aimed at improving drug use and patient safety. It includes a finished analysis of the therapy indicated by the physician, evaluating the safer alternatives for the type of patient and the special conditions of his pathology, emphasizing evaluations of the effectiveness, safety and tolerability of the medication, drug interactions, possible events Adverse effects, dose adjustments by sea, patient conditions; Verification of what the sea of optimal management, including the choice of the best route for the shelf and the time in which the medicines are infused to the patient.

The intervention is performed at moments one during the stay in the service where they communicate and educate the patient about all the medications indicated and the relationship, which have their health status, as well as the benefits and expected results with their administration. A second moment just after high medicine, where the same review of medications is done and recommendations are given to the patient on how to administer them, promoting adherence to treatment. In addition to all the knowledge he has about his pathology and treatment.

To see that the patient started therapy, the last 7 days after discharge / transfer of the Emergency Service, a member of the team communicated by telephone with the patient. In case you have not started looking for the factors that affected your behavior.

At 30 days after discharge / transfer, an independent external evaluator, blinded to pharmaceutical care, who will not know the group to which the patient belongs, will be contacted by telephone and evaluated again, in addition to consulting medical prescriptions Received and medications purchased to evaluate hospital readmissions or unscheduled medical consultations.

If an error is detected in the control group, it will be communicated to the health team

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department of clinical hospital of the University of Chile
* Patients who sign the informed consent form
* Patients in triage categories C2, C3, C4 and C5

Exclusion Criteria:

* Patients with inability to communicate and don't have a responsible caregiver to provide reliable information about the patient's therapy
* Patients who are participating in another study
* Patients not taking drugs regularly and who don't receive them during care in the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
User satisfaction | 4 months

SECONDARY OUTCOMES:
Readmission | 4 months
Drug Related Problem | 4 months
Adherence measured by four question Morisky-Green test | 5 months
  If the patient answers all question "NO", the patient is adherent. Measured in two times in the study. The proportion of adherent patients will be measured with respect to the total of them.
Proportion of recommendations to the health team accepted | 4 months
  Recommendations made by a clinical pharmacist can be accepted or rejected. The measurement will be (accepted recommendations/total of recommendations) x100

CONTACTS AND LOCATIONS:
Overall Officials: Matías Martínez, Msc, Principal Investigator — University of Chile

IPD SHARING:
Plan to Share IPD: No